CLINICAL TRIAL: NCT01275144
Title: Effect of LY2216684 on the Pharmacokinetics and Pharmacodynamics of Lorazepam in Healthy Subjects
Brief Title: A Study of the Effect of LY2216684 on Lorazepam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12596; H9P-EW-LNCG (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2216684+lorazepam, placebo+lorazepam (Experimental): Oral 18 mg doses of LY2216684 on days 1-6 with a single oral 1 mg dose of lorazepam on day 3 in treatment period 1. Oral doses of placebo on days 1-6 with a single oral 1 mg dose of lorazepam on day 3 in treatment period 2. There is a washout period of at least 7 days between dosing periods.
  Interventions: Drug: LY2216684; Drug: Placebo; Drug: Lorazepam
- Placebo+Lorazepam, LY2216684+Lorazepam (Experimental): Oral doses of placebo on days 1-6 with a single oral 1 mg dose of lorazepam on day 3 in treatment period 1. Oral 18 mg doses of LY2216684 on days 1-6 with a single oral 1 mg dose of lorazepam on day 3 in treatment period 2. There is a washout period of at least 7 days between dosing periods.
  Interventions: Drug: LY2216684; Drug: Placebo; Drug: Lorazepam

INTERVENTIONS:
Drug: LY2216684 — Administered orally
Drug: Placebo — Administered orally
Drug: Lorazepam — Administered orally

SUMMARY:
The purpose of this study is to determine how much lorazepam gets into the blood and how long it takes the body to get rid of it when given together with LY2216684. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy, as determined by medical history and physical examination.
* Male participants - Agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.
* Female participants - Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug; or Women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone [FSH] >40 milli-international Units per milliliter [mIU/mL]).
* Have a body weight >50 kilogram (kg).
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator (potassium, magnesium, and calcium values must be within the normal range).
* Have venous access sufficient to allow blood sampling as per the protocol.
* Have normal blood pressure and pulse rate (sitting position) as determined by the investigator.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device other than the study drug, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2216684, lorazepam, benzodiazepines, or related compounds.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to screening.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have a history or show evidence of significant active neuropsychiatric disease or have a history of suicide attempt or ideation.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Intend to use over-the-counter or prescription medication (including hormonal contraceptives) within 14 days prior to dosing unless deemed acceptable by the investigator and Sponsor's medical monitor, except for influenza vaccinations.
* Use of any drugs or substances that are known to be substrates, inducers, or inhibitors of Uridine 5'-diphospho -glucuronosyltransferase (UGT) within 30 days prior to dosing.
* Have donated blood of more than 500 mL within the last month.
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption 48 hours prior to each study period and while resident at the clinical research unit (CRU) (1 unit = 12 ounces (oz) or 360 millimeters (mL) of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participants unwilling to adhere to study caffeine restrictions.
* Have used any tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment and during the study.
* Have a documented or suspected history of acute narrow angle glaucoma.
* Have Gilbert's Syndrome
* Participants determined to be unsuitable by the investigator for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Leeds, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2216684 + Lorazepam, Then Placebo + Lorazepam: Period 1, 18 milligram (mg) dose of LY2216684 on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3. Period 2, dose of Placebo on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3.
- Placebo + Lorazepam, Then LY2216684 + Lorazepam: Period 1, dose of Placebo on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3.Period 2, 18 milligram (mg) dose of LY2216684 on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3.
Period: First Intervention (6 Days)
Arm/Group | LY2216684 + Lorazepam, Then Placebo + Lorazepam | Placebo + Lorazepam, Then LY2216684 + Lorazepam
Started | 14 | 14
Received at Least 1 Dose of Study Drug | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | LY2216684 + Lorazepam, Then Placebo + Lorazepam | Placebo + Lorazepam, Then LY2216684 + Lorazepam
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Second Intervention (6 Days)
Arm/Group | LY2216684 + Lorazepam, Then Placebo + Lorazepam | Placebo + Lorazepam, Then LY2216684 + Lorazepam
Started | 14 | 14
Completed | 13 | 14
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: All randomized participants
Arm/Group | Overall
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Black or African American | 5
  Multiple | 4
  White | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Lorazepam, Maximum Plasma Concentration (Cmax)
Description: The geometric least squares mean and 90% Confidence Interval are presented. Geometric least squares mean corrected for participant, treatment and random error.
Time Frame: Predose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post lorazepam dose
Population: All enrolled participants.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Groups:
- LY2216684 + Lorazepam: Oral 18 mg dose of LY2216684 on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3
- Placebo + Lorazepam: Oral dose of Placebo on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
nanograms per milliliter (ng/mL) | 9.620 [9.178 to 10.083] | 10.720 [10.228 to 11.236]
Statistical Analysis 1: Comparison: LY2216684 + Lorazepam vs Placebo + Lorazepam; Test type: Superiority or Other; Ratio of geometric least square mean = 0.897, 90% CI 2-sided [0.86 to 0.94] — Ratio of LY2216684 to Placebo

2. Primary Outcome: Pharmacokinetics of Lorazepam, Time to Maximum Plasma Concentration (Tmax)
Time Frame: Predose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post lorazepam dose
Population: All enrolled participants
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
hours | 3.00 [1.08 to 4.02] | 2.00 [1.00 to 4.00]
Statistical Analysis 1: Comparison: LY2216684 + Lorazepam vs Placebo + Lorazepam; Test type: Superiority or Other; p = 0.0021, Wilcoxon signed rank test; median of paired differences = 0.50, 90% CI 2-sided [0.50 to 1.00] — Ratio of LY2216684 to Placebo

3. Primary Outcome: Pharmacokinetics of Lorazepam, Area Under the Plasma Concentration Curve (AUC) From Time 0 to Infinity (∞)
Description: as for outcome 1
Time Frame: Predose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post lorazepam dose
Population: All enrolled participants
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
nanograms*hour per milliliter (ng*h/mL) | 207 [193 to 222] | 199 [185 to 213]
Statistical Analysis 1: Comparison: LY2216684 + Lorazepam vs Placebo + Lorazepam; Test type: Superiority or Other; Ratio of geometric least square mean = 1.04, 90% CI 2-sided [1.01 to 1.08] — Ratio of LY2216684 to Placebo

4. Secondary Outcome: Change From Baseline in Cognitive Function-Simple Reaction Time
Description: Participants were instructed to press the 'Yes' response button as quickly as possible every time the word 'Yes' was presented on the computer screen. Fifty stimuli were presented with a varying inter-stimulus interval of between 1 and 3.5 seconds. Participant's reaction time to the stimulus was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: millisecond (msec)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
millisecond (msec)
  Day 3, 2 hours | 5.0102 (8.8823) | 23.9962 (8.8823)
  Day 3, 4 hours | 27.9731 (8.8823) | 40.0858 (8.8823)
  Day 3, 8 hours | 13.1424 (8.8823) | 10.0183 (8.8823)

5. Secondary Outcome: Change From Baseline in Cognitive Function-Digit Vigilance Targets Detected
Description: A target digit was pseudo-randomly selected and constantly displayed to the right of the computer screen. A series of 450 digits was then presented in the center of the computer screen at the rate of 150 per minute. The participant was required to press the 'Yes' button as quickly as possible every time a digit in the series matched the target digit. There were 45 targets. Percentage of target digits correctly detected was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: percentage of digits correctly detected
Units Other Than Participants: Obsevations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (Obsevations) | 56 | 56
percentage of digits correctly detected
  Day 3, 2 hours | -3.5852 (1.3892) | -3.5577 (1.3892)
  Day 3, 4 hours | -2.4745 (1.3892) | -4.1927 (1.3892)
  Day 3, 8 hours | -2.5534 (1.3892) | -1.9702 (1.3892)

6. Secondary Outcome: Change From Baseline in Cognitive Function-Digit Vigilance Speed
Description: A target digit was pseudo-randomly selected and constantly displayed to the right of the computer screen. A series of 450 digits was then presented in the center of the computer screen at the rate of 150 per minute. The participant was required to press the 'Yes' button as quickly as possible every time a digit in the series matched the target digit. There were 45 targets. Speed at which a participant detected target digits was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: millisecond (msec)
Units Other Than Participants: Observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (Observations) | 56 | 56
millisecond (msec)
  Day 3, 2 hours | 20.1712 (7.0627) | 12.0238 (7.0627)
  Day 3, 4 hours | 14.7702 (7.0627) | 12.1391 (7.0627)
  Day 3, 8 hours | 9.8277 (7.0627) | 2.5073 (7.0627)

7. Secondary Outcome: Change From Baseline in Cognitive Function-Digit False Alarms
Description: A target digit was pseudo-randomly selected and constantly displayed to the right of the computer screen. A series of digits were then presented in the center of the computer screen at the rate of 150 per minute. The participant was required to press the 'Yes' button as quickly as possible every time a digit in the series matched the target digit. There were 45 targets. The number of false alarms (incorrect 'Yes' responses) was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: Number of false alarms
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
Number of false alarms
  Day 3, 2 hours | 1.0204 (0.3122) | 0.7296 (0.3122)
  Day 3, 4 hours | 0.1990 (0.3122) | 1.0510 (0.3122)
  Day 3, 8 hours | 0.4490 (0.3122) | 0.7653 (0.3122)

8. Secondary Outcome: Change From Baseline in Cognitive Function-Choice Reaction Time
Description: Participants were required to respond to the words 'Yes' and 'No' as they appeared on the computer screen by pressing the corresponding button as quickly as possible. There were 50 trials during which each stimulus word was chosen randomly with equal probability; there was a varying inter-stimulus interval of between 1 and 3.5 seconds. The time required to respond was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: millisecond (msec)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
millisecond (msec)
  Day 3, 2 hours | 28.2448 (12.6614) | 8.4745 (12.6614)
  Day 3, 4 hours | 8.9837 (12.6614) | 10.6866 (12.6614)
  Day 3, 8 hours | 9.7930 (12.6614) | -13.1780 (12.6614)

9. Secondary Outcome: Change From Baseline in Cognitive Function-Choice Reaction Time Accuracy
Description: Participants were required to respond to the words 'Yes' and 'No' as they appeared on the computer screen by pressing the corresponding button as quickly as possible. There were 50 trials during which each stimulus word was chosen randomly with equal probability; there was a varying inter-stimulus interval of between 1 and 3.5 seconds. The percentage of correct responses was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: percentage of correct responses
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
percentage of correct responses
  Day 3, 2 hours | -1.2292 (0.7353) | -0.4851 (0.7353)
  Day 3, 4 hours | -1.3720 (0.7353) | -1.2708 (0.7353)
  Day 3, 8 hours | -0.5863 (0.7353) | -1.1994 (0.7353)

10. Secondary Outcome: Change From Baseline in Cognitive Function-Numeric Working Memory Sensitivity Index (SI)
Description: Working memory is a sum of accuracy measures from the numeric and spatial working memory tasks (sensitivity index [SI]). Working Memory SI is based on how fast the participant responds correctly and how many are correct responses. A high score reflects someone able to hold in memory for a prolonged period. A negative change from baseline reflects impairment compared to baseline.
  A series of 5 digits were presented on a computer screen, one every 1.15 seconds, for the participant to hold in memory. This was followed by a series of 30 probe digits for each of which the participant had to decide whether it had appeared in the original series of digits and press the corresponding 'Yes' or 'No' response button as quickly as possible. This procedure was repeated 2 times using 2 different series and probes. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: Sensitivity Index (SI)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
Sensitivity Index (SI)
  Day 3, 2 hours | -0.00764 (0.02639) | 0.003388 (0.02639)
  Day 3, 4 hours | -0.02121 (0.02639) | -0.00511 (0.02639)
  Day 3, 8 hours | 0.007112 (0.02639) | -0.01865 (0.02639)

11. Secondary Outcome: Change From Baseline in Cognitive Function-Numeric Working Memory Speed
Description: A series of 5 digits were presented on a computer screen, one every 1.15 seconds, for the participant to hold in memory. This was followed by a series of 30 probe digits for each of which the participant had to decide whether it had appeared in the original series of digits and press the corresponding 'Yes' or 'No' response button as quickly as possible. This procedure was repeated a further 2 times using 2 different series and probes. The time required to press the corresponding 'Yes' or 'No' response button in response to the probe digit is presented. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
milliseconds (msec)
  Day 3, 2 hours | 58.2923 (27.7074) | 72.0037 (27.7074)
  Day 3, 4 hours | 8.1891 (27.7074) | 25.5894 (27.7074)
  Day 3, 8 hours | -33.6927 (27.7074) | -14.5106 (27.7074)

12. Secondary Outcome: Change From Baseline in Cognitive Function-Immediate Word Recall Accuracy
Description: The participant was given a series of words to commit to memory. Immediately after the last word was presented, the participant was given 1 minute to write as many of the words as possible in any order on a sheet of paper. The percentage of words correctly recalled (present on the original list of words) was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: percentage of words correctly recalled
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
percentage of words correctly recalled
  Day 3, 2 hours | -2.2751 (1.8276) | -3.6767 (1.8276)
  Day 3, 4 hours | -7.2744 (1.8276) | -5.8195 (1.8276)
  Day 3, 8 hours | -4.4166 (1.8276) | -4.1524 (1.8276)

13. Secondary Outcome: Change From Baseline in Cognitive Function-Immediate Word Recall Errors
Description: The participant was given a series of words to commit to memory. Immediately after the last word was presented, the participant was given 1 minute to write as many of the words as possible in any order on a sheet of paper. The number of words incorrectly recalled (not on the original list of words) was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: number of words incorrectly recalled
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
number of words incorrectly recalled
  Day 3, 2 hours | -0.1582 (0.1494) | 0.1225 (0.1494)
  Day 3, 4 hours | 0.05605 (0.1494) | 0.2297 (0.1494)
  Day 3, 8 hours | 0.05605 (0.1494) | 0.3011 (0.1494)

14. Secondary Outcome: Change From Baseline in Cognitive Function-Delayed Word Recall Accuracy
Description: The participant was given a series of words to commit to memory. After a delay of approximately 15-20 minutes, the participant was given 1 minute to write as many of the words as possible in any order on a sheet of paper. The percentage of words correctly recalled (present on the original list of words) was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: percentage of words correctly recalled
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
percentage of words correctly recalled
  Day 3, 2 hours | -2.0338 (1.8465) | -6.2980 (1.8465)
  Day 3, 4 hours | -10.8423 (1.8465) | -8.2034 (1.8465)
  Day 3, 8 hours | -11.5566 (1.8465) | -6.0595 (1.8465)

15. Secondary Outcome: Change From Baseline in Cognitive Function-Delayed Word Recall Errors
Description: The participant was given a series of words to commit to memory. After a delay, the participant was given 1 minute to write as many of the words as possible in any order on a sheet of paper. The number of incorrect words was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: number of words incorrectly recalled
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
number of words incorrectly recalled
  Day 3, 2 hours | 0.1535 (0.2448) | 0.6323 (0.2448)
  Day 3, 4 hours | 0.6535 (0.2448) | 0.8108 (0.2448)
  Day 3, 8 hours | 0.6177 (0.2448) | 0.4180 (0.2448)

16. Secondary Outcome: Change From Baseline in Cognitive Function-Word Recognition Sensitivity Index (SI)
Description: Word Recognition SI is based on how fast the participant responds correctly and how many are correct responses. SI ranging from zero (chance performance) to one (perfect accuracy). Higher SI indicates better cognitive function. A negative change from baseline reflects impairment compared to baseline.
  The original words from Word Presentation plus 15 distractor words were presented one at a time in a randomized order. For each word, the participant was required to indicate whether they recognized it from the original list of words by pressing the corresponding 'Yes' or 'No' button as quickly as possible. Following each response, there was a delay of 1 second before the next word was presented. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: Sensitivity Index (SI)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
Sensitivity Index (SI)
  Day 3, 2 hours | -0.08834 (0.04199) | -0.07719 (0.04199)
  Day 3, 4 hours | -0.06242 (0.04199) | -0.1983 (0.04199)
  Day 3, 8 hours | -0.1523 (0.04199) | -0.1524 (0.04199)

17. Secondary Outcome: Change From Baseline in Cognitive Function-Word Recognition Speed
Description: The original words from Word Presentation plus 15 distractor words were presented one at a time in a randomized order. For each word, the participant was required to indicate whether they recognized it from the original list of words by pressing the corresponding 'Yes' or 'No' button as quickly as possible. Following each response, there was a delay of 1 second before the next word was presented. The time required to press the corresponding 'Yes' or 'No' response button in response to the word was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
milliseconds (msec)
  Day 3, 2 hours | -13.7645 (36.5329) | -6.3483 (36.5329)
  Day 3, 4 hours | -39.5052 (36.5329) | -25.9919 (36.5329)
  Day 3, 8 hours | -40.9574 (36.5329) | -133.24 (36.5329)

18. Secondary Outcome: Change From Baseline in Cognitive Function-Picture Recognition Sensitivity Index (SI)
Description: Picture Recognition SI is based on how fast the participant responds correctly and how many are correct responses. SI ranging from zero (chance performance) to one (perfect accuracy). Higher SI indicates better cognitive function. A negative change from baseline reflects impairment compared to baseline.
  The original pictures from Picture Presentation plus 20 distractor pictures were presented one at a time. For each picture, the participant was required to indicate whether they recognized it from the original series of pictures by pressing the corresponding 'Yes' or 'No' button as quickly as possible. Following the response, there was a delay of 1 second before the next pictures was presented. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: Sensitivity Index
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
Sensitivity Index
  Day 3, 2 hours | 0.02080 (0.04778) | -0.03440 (0.04778)
  Day 3, 4 hours | -0.04431 (0.04778) | -0.06015 (0.04778)
  Day 3, 8 hours | -0.1054 (0.04778) | -0.09855 (0.04778)

19. Secondary Outcome: Change From Baseline in Cognitive Function-Picture Recognition Speed
Description: The original pictures from Picture Presentation plus 20 distractor pictures were presented one at a time. For each picture, the participant was required to indicate whether they recognized it from the original series of pictures by pressing the corresponding 'Yes' or 'No' button as quickly as possible. Following the response, there was a delay of 1 second before the next pictures was presented. The time required to press the corresponding 'Yes' or 'No' response button in response to the picture was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
milliseconds (msec)
  Day 3, 2 hours | 57.2341 (37.5217) | 144.67 (37.5217)
  Day 3, 4 hours | 51.7809 (37.5217) | 62.2059 (37.5217)
  Day 3, 8 hours | -59.9669 (37.5217) | -23.2941 (37.5217)

20. Secondary Outcome: Change From Baseline in Cognitive Function-Tracking Average Distance From Target
Description: The participant used a joystick to track a randomly moving target on the computer screen. The distance from the target was measured. Participant's response was measured twice. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
millimeters (mm)
  Day 3, 2 hours | 0.3850 (2.4910) | -0.3614 (2.4910)
  Day 3, 4 hours | 6.1672 (2.4910) | -0.1104 (2.4910)
  Day 3, 8 hours | 0.3743 (2.4910) | -0.6036 (2.4910)

21. Secondary Outcome: Change From Baseline in Cognitive Function-Postural Stability
Description: The ability to stand upright without moving was assessed using equipment modeled on the Wright Ataxia-meter. To measure movements, a cord was attached to the participant who was required to stand for one minute, as still as possible, with feet apart and eyes closed. The amount of sway is expressed as the total angular movement calibrated in units of one-third degree of angle of sway.
  The amount of sway is expressed as the total angular movement in the antero-posterior plane and calibrated in units of one-third degree of angle of sway. Higher result indicates better postural stability. A negative change from baseline reflects impairment compared to baseline. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: 1/3 degree of angle of sway
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
1/3 degree of angle of sway
  Day 3, 2 hours | -1.5464 (2.0012) | 9.1392 (2.0012)
  Day 3, 4 hours | 0.1965 (2.0012) | 2.1857 (2.0012)
  Day 3, 8 hours | -0.9571 (2.0012) | -1.6429 (2.0012)

22. Secondary Outcome: Change From Baseline in Cognitive Function-Self-rated Alertness
Description: The participant was required to rate how they felt "at this moment" on sixteen 10 centimeter visual analogue scales. The scale endpoints were anchored using polar word pairs such as 'drowsy-alert', 'clumsy-well coordinated', 'mentally slow-quick witted' and 'incompetent-proficient'. Responses from the 16 scales were scored to yield 3 main factors: Self-rated Alertness, Self-rated Contentment, and Self-rated Calmness. The possible range of scores are 0 to 100 for each factor and are represented in millimeters on the 10 centimeter line with higher numbers indicating greater alertness. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
millimeters (mm)
  Day 3, 2 hours | 5.1411 (2.4896) | 3.2597 (2.4896)
  Day 3, 4 hours | 3.6887 (2.4896) | 4.0018 (2.4896)
  Day 3, 8 hours | 3.7205 (2.4896) | 3.1287 (2.4896)

23. Secondary Outcome: Change From Baseline in Cognitive Function-Self-rated Contentment
Description: The participant was required to rate how they felt "at this moment" on sixteen 10 centimeter visual analogue scales. The scale endpoints were anchored using polar word pairs such as 'drowsy-alert', 'clumsy-well coordinated', 'mentally slow-quick witted' and 'incompetent-proficient'. Responses from the 16 scales were scored to yield 3 main factors: Self-rated Alertness, Self-rated Contentment, and Self-rated Calmness. The possible range of scores are 0 to 100 for each factor and are represented in millimeters on the 10 centimeter line with higher numbers indicating greater contentment. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
millimeters (mm)
  Day 3, 2 hours | 3.1100 (1.9527) | 1.3686 (1.9527)
  Day 3, 4 hours | 3.0171 (1.9527) | 3.3829 (1.9527)
  Day 3, 8 hours | 3.3743 (1.9527) | 0.01857 (1.9527)

24. Secondary Outcome: Change From Baseline in Cognitive Function-Self-rated Calmness
Description: The participant was required to rate how they felt "at this moment" on sixteen 10 centimeter visual analogue scales. The scale endpoints were anchored using polar word pairs such as 'drowsy-alert', 'clumsy-well coordinated', 'mentally slow-quick witted' and 'incompetent-proficient'. Responses from the 16 scales were scored to yield 3 main factors: Self-rated Alertness, Self-rated Contentment, and Self-rated Calmness. The possible range of scores are 0 to 100 for each factor and are represented in millimeters on the 10 centimeter line with higher numbers indicating greater calmness. Least squares means were adjusted for baseline, period, sequence, time, treatment and treatment*time.
Time Frame: Baseline, 2, 4, 8 hours on Day 3
Population: All enrolled participants
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Units Other Than Participants: observations
Arm/Group | LY2216684 + Lorazepam | Placebo + Lorazepam
Number analyzed (Participants) | 28 | 28
Number analyzed (observations) | 56 | 56
millimeters (mm)
  Day 3, 2 hours | -0.9651 (1.9110) | 0.3401 (1.9110)
  Day 3, 4 hours | 1.4099 (1.9110) | -1.3564 (1.9110)
  Day 3, 8 hours | 3.4635 (1.9110) | 0.3936 (1.9110)

ADVERSE EVENTS:
Groups:
- LY2216684: Oral 18 mg dose of LY2216684 on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3; Serious and Other Adverse Events assessed on Days 1 and 2
- Placebo: Oral dose of Placebo on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3; Serious and Other Adverse Events assessed on Days 1 and 2
- LY2216684 + Lorazepam: Oral 18 mg dose of LY2216684 on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3; Serious and Other Adverse Events assessed on Days 3-6
- Placebo + Lorazepam: Oral dose of Placebo on Days 1-6 with a single oral 1 mg dose of lorazepam on Day 3; Serious and Other Adverse Events assessed on Days 3-6
Arm/Group | LY2216684 | Placebo | LY2216684 + Lorazepam | Placebo + Lorazepam
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 13/28 | 3/28 | 6/28 | 4/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 (N=28) | Placebo (N=28) | LY2216684 + Lorazepam (N=28) | Placebo + Lorazepam (N=28)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Semenuria (Renal and urinary disorders) | 0/23 (0) | 0/23 (0) | 1/23 (1) | 0/23 (0)
Urinary hesitation (Renal and urinary disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 0/23 (0) | 0/23 (0) | 1/23 (1) | 0/23 (0)
Penis disorder (Reproductive system and breast disorders) | 0/23 (0) | 0/23 (0) | 1/23 (1) | 0/23 (0)
Scrotal pain (Reproductive system and breast disorders) | 0/23 (0) | 0/23 (0) | 1/23 (1) | 0/23 (0)
Testicular pain (Reproductive system and breast disorders) | 0/23 (0) | 0/23 (0) | 1/23 (1) | 0/23 (0)
Testicular retraction (Reproductive system and breast disorders) | 1/23 (1) | 0/23 (0) | 0/23 (0) | 0/23 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days